CLINICAL TRIAL: NCT05098379
Title: A Tele-Rehabilitation Home Exercise Program to Promote Fitness and Functional Mobility in Ambulatory Adults With Cerebral Palsy: A Feasibility Study
Brief Title: Tele-Rehabilitation Home Exercise Program for Ambulatory Adults With Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAAT5675
Record Dates: First submitted 2021-10-15; First posted 2021-10-28 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Cerebral Palsy
Keywords: Exercise; Telehealth; Rehabilitation
MeSH Terms: conditions — Cerebral Palsy; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tele-Rehabilitation Home Exercise Program (Experimental): Subjects will participate in an 8-week customized home exercise program with weekly virtual exercise coaching sessions.
  Interventions: Behavioral: Tele-Rehabilitation Home Exercise Program

INTERVENTIONS:
Behavioral: Tele-Rehabilitation Home Exercise Program — Participants will engage in 150 minutes of exercise per week (30 min/day for 5 days/week) for 8 weeks and will have weekly virtual Exercise Coaching sessions with a trained project team member. Customized home exercise programs will be reviewed weekly during the coaching sessions and will be modified as needed to ensure participants can complete their exercises safely and effectively. Exercise coaches will send weekly messages to 'check-in' with participants in order to motivate and remind participants to adhere to their tailored home exercise programs.
  During weekly exercise coaching sessions, exercises will be reviewed for form, safety, and progression. Exercises will be revised as needed to ensure that they are in line with participants' goals, needs, and preferences.

SUMMARY:
This study aims to determine if a tele-rehabilitation home exercise program is feasible to promote adherence to a fitness and mobility exercise program in ambulatory adults with cerebral palsy (GMFCS I, II, III) aged 21- 60 year old, and second, to determine if a tele-health exercise program improves fitness and functional mobility for participants.

DETAILED DESCRIPTION:
Cerebral palsy (CP) is a non-progressive neurologic condition caused by a brain lesion(s) that occurs in the prenatal, perinatal or early postnatal period. Ambulatory adults with CP are at risk for gait deterioration and increased sedentary lifestyles due to their diagnosis, associated conditions and the impact of aging. Adults with CP often have limited access to physical therapy (PT) and community-based programs to sustain ambulation, reduce pain, prevent falls risk and increase fitness and physical activity. This Tele-Rehabilitation Home Exercise Program (TRHExP) is a prospective cohort study

Participants in this feasibility study will engage in 150 minutes of exercise per week (30 min/day for 5 days/week) for 8 weeks and will have weekly virtual Exercise Coaching sessions with a trained project team member.

ELIGIBILITY:
Inclusion Criteria:

* Primary diagnosis: Spastic Cerebral Palsy (unilateral or bilateral)
* Gross Motor Function Classification System (GMFCS) Level I to III
* No orthopedic surgery in past year
* No Botox in past 3 months
* Able to follow directions & attend for 20-30 minutes
* Able to stand independently up to 1 minutes with or without an assistive device
* Able to walk independently up to 2 minutes with or without an assistive device
* Must have a laptop, tablet or smart phone to do the program

Exclusion Criteria:

* Visual, cognitive or attentional deficit that makes it too difficult to participate
* No technology to participate in Zoom tele-rehabilitation sessions
* Medical contraindications to participate in an Exercise Program (e.g., uncontrolled hypertension, diabetes, syncope, uncontrolled seizures)

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2021-10-31 (Actual); Primary Completion 2022-05-08 (Actual); Study Completion 2022-05-08 (Actual)

PRIMARY OUTCOMES:
Canadian Occupational Performance Measure (COPM) | Baseline
  The COPM is a semi-structured interview that measures participants' perspective of their performance and satisfaction of self-identified occupational performance problems in areas of self-care, productivity and leisure. Participants rate their performance and satisfaction of the occupational performance problems they identify using a 10 point scale. Scores range from 1 to 10, with 1 indicating poor performance/ low satisfaction and 10 indicating very good performance/ high satisfaction (better outcome).
Canadian Occupational Performance Measure (COPM) | 8 weeks (Post-Test)
  The COPM is a semi-structured interview that measures participants' perspective of their performance and satisfaction of self-identified occupational performance problems in areas of self-care, productivity and leisure. Participants rate their performance and satisfaction of the occupational performance problems they identify using a 10 point scale. Scores range from 1 to 10, with 1 indicating poor performance/ low satisfaction and 10 indicating very good performance/ high satisfaction (better outcome).

SECONDARY OUTCOMES:
30 Second Sit to Stand Test | Baseline, 8 weeks (Post-Test)
  The participant is asked to stand up from a standard chair without using their arms as many times as possible within 30 seconds. The number of full stands are counted.
2 Minute Step Test | Baseline, 8 weeks (Post-Test)
  The participant is asked to stand next to the wall, and a piece of tape is placed on the wall halfway between the participant's iliac crest and patella. The participant is asked to step in place for 2 minutes, raising each knee to the mark on the wall for each step, for as many times as possible within that period. The number of times the right knee reaches the required height are counted.
Single Leg Stance Measure | Baseline, 8 weeks (Post-Test)
  The participant is asked to stand unassisted on one leg with eyes open and hands on hips. The amount of time in seconds the participant can maintain this position is measured (up to 30 seconds).
Patient-Reported Outcomes Measurement Information Systems (PROMIS) Pediatric Short Form (SF) v1.0 - Physical Activity 4a | Baseline, 8 weeks (Post-Test)
  This is a 4-item questionnaire that asks participants about their level of physical activity in the past 7 days. Items are scored on a 5-point scale. Scores range from 4 to 20 with 4 indicating low physical activity and 20 indicating high physical activity (better outcome).
PROMIS SF v2.0 - Physical Function 10a | Baseline, 8 weeks (Post-Test)
  This is a 10-item questionnaire that asks participants about their level of physical function. Items are scored on a 5-point scale. Scores range from 10 to 50 with 10 indicating high physical function (better outcome) and 50 indicating low physical function.
PROMIS Scale v2.0 - Pain Intensity 3a | Baseline, 8 weeks (Post-Test)
  This is a 3-item questionnaire that asks participants about their pain intensity. Items are scored on a 5-point scale. Scores range from 3 to 15 with 3 indicating "no pain" (better outcome) and 15 indicating "very severe pain".
PROMIS SF v1.1-Pain Interference 8a | Baseline, 8 weeks (Post-Test)
  This is an 8-item questionnaire that asks participants about how much pain interferes with daily life. Items are scored on a 5-point scale. Scores range from 8 to 40, with 8 indicating "not at all" (better outcome) and 40 indicating "very much".
PROMIS SF v1.0 - Fatigue 8a | Baseline, 8 weeks (Post-Test)
  This is an 8-item questionnaire that asks participants about how much they were affected by fatigue in the past 7 days. Items are scored on a 5-point scale.
  Score range from 8-40 with 8 indicating "not at all" (better outcome) and 40 indicating "very much".

CONTACTS AND LOCATIONS:
Overall Officials: Joel Stein, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

REFERENCES:
- [Background] Rosenbaum P, Paneth N, Leviton A, Goldstein M, Bax M, Damiano D, Dan B, Jacobsson B. A report: the definition and classification of cerebral palsy April 2006. Dev Med Child Neurol Suppl. 2007 Feb;109:8-14. PMID 17370477
- [Background] Turk MA. Health, mortality, and wellness issues in adults with cerebral palsy. Dev Med Child Neurol. 2009 Oct;51 Suppl 4:24-9. doi: 10.1111/j.1469-8749.2009.03429.x. PMID 19740207
- [Background] Rimmer JH, Riley B, Wang E, Rauworth A, Jurkowski J. Physical activity participation among persons with disabilities: barriers and facilitators. Am J Prev Med. 2004 Jun;26(5):419-25. doi: 10.1016/j.amepre.2004.02.002. PMID 15165658